CLINICAL TRIAL: NCT03391557
Title: Significance of Endoscopic Ultrasonography Guided Transbronchial Lymph Node Biopsy (TBNA) and Ultrasound Elastography in Lymph Node
Brief Title: Significance of Ultrasound Elastography in Lymph Node
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fangsurong (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Fangsurong, Deputy chief physician, master, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YL20160713-020
Record Dates: First submitted 2017-12-23; First posted 2018-01-05 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: Elastography; Lymph node; Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Patients who underwent EBUS-TBNA examination in department of respiration,Nanjing Hospital Affiliated to Nanjing Medical University during 21June 2016 and 17 April 2017 were included in the study, All patients were evaluated by chest enhanced CT and/or 18-FDG PET-CT,those who had enlarged intrathoracic lymph nodes(≥1cm) and/or 18-FDG high uptake (SUV Max > 2.5) without bleeding tendency, abnormal coagulation function and serious cardiac dysfunction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with the UE examination (Experimental): Patients with enlarged intrathoracic lymph nodes(≥1cm) and/or 18-FDG high uptake (SUV Max > 2.5) without bleeding tendency, abnormal coagulation function and serious cardiac dysfunction were finally selected.
  Interventions: Diagnostic Test: UE

INTERVENTIONS:
Diagnostic Test: UE — All patients were examined by enhanced chest computed tomography (CT), the B-mode ultrasound and endobronchial ultrasound (EBUS)guided elastography before EBUS-TBNA. Each lymph node was assessed by describing the characteristics of the CT image (short diameter, texture, shape, boundary, mean CT value), B-mode ultrasound (short diameter, echo characteristic, shape, boundary) and ultrasound elastography (image type, grading score, strain rate, blue area ratio).
  Other Names: Ultrasound Elastography

SUMMARY:
Background and Objectives: Elastography can reflect the difference of tissue hardness, which helps to identify the difference of hardness between benign and malignant tissues. The aim of this study was to evaluate the value of endobronchial ultrasound elastography in the differential diagnosis of benign and malignant intrathoracic lymph nodes. Materials and Methods: A total of 42 patients with intrathoracic lymphadenopathy required for EBUS-TBNA examination were prospectively enrolled. Firstly, All patients were evaluated by enhanced chest CT examination,the EBUS B-mode ultrasound and EBUS-guided elastography before EBUS-TBNA.Then, the investigators evaluated every lymph node by describing the characteristics of the CT image (Short diameter, texture, shape, boundary ,mean CT value), B-mode ultrasound (short diameter, echo characteristic, shape, boundary) and elastography (image type, grading score, strain rate, blue area ratio). Finally, the pathological results were used as the gold standard. the investigators compare the characteristics of the 3 evaluating methods alone and in combination between benign and malignant lymph nodes.

DETAILED DESCRIPTION:
Introduction Elastography was first proposed by Ophir of Texas State University in the United States in 1991 ，which can objectively reflect the elastic information of the tissue through the deformation of the external force. Then, the elastic information is converted to RGB (red,green,blue) mode image, where hard tissue is shown in blue, medium tissue in green and soft tissue in red, overlaid on the B-mode image. Different image colors reflect the difference of tissue hardness, and then help identify the difference between benign and malignant tissue hardness. UE has become a hot spot in medical ultrasound imaging shortly after it was proposed. Now UE is widely used in the diagnosis of diseases in the breast, thyroid, prostate and other related tissues. The common clinical UE includes quasi-static elasiticity imaging, acoustic radiation force pulse (ARFI) and shear wave elastography (SWE).

Lung cancer is one of the most common malignancies with high morbidity and mortality，the 5-year survival rate being only 16%. Lymphatic metastasis, the most common mode of metastasis, is of great significance for staging of lung cancer. Therefore, the correct diagnosis of benign and malignant intrathoracic lymph nodes becomes the key to definite diagnosis and accurate treatment. EBUS-TBNA has shown its certain diagnostic value in lung cancer, lymphoma, sarcoidosis and lymph node tuberculosis. However, researches related to real-time endobronchial UE (EBUS-RTE) are scarce, EBUS-RTE combined with EBUS B-mode ultrasound and enhanced CT is even fewer.

This study aimed to evaluate the value of endobronchial UE in differentiating benign and malignant intrathoracic lymph nodes qualitatively and quantitatively, and the combined features were evaluated as well. Here we show that endobronchial UE has significant value in the differential diagnosis of benign and malignant intrathoracic lymph nodes.

Materials and Methods Patients Patients undergoing EBUS-TBNA examination in the Department of Respiratory Diseases, Nanjing Hospital Affiliated to Nanjing Medical University from June 2016 to April 2017 were recruited in this study. All patients were evaluated by chest enhanced CT and/or 18-FDG PET-CT. Those who had enlarged intrathoracic lymph nodes(≥1cm) and/or 18-FDG high uptake (SUV Max > 2.5) without bleeding tendency, abnormal coagulation function and serious cardiac dysfunction were finally selected. The study was approved by the Ethics Committee of Nanjing Hospital (YL 20160713-020) and supported by Nanjing Science and Technology Commission (201505002). All the patients gave written informed consent.

EBUS B-Mode ultrasound The patients were sedated by local anesthesia (lidocaine, China Otsuka Pharmaceutical Incorporated Company) and conscious sedation (midazolam, Jiangsu Nhwa Pharmaceutical incorporated company; fentanyl, Yichang Humanwell Pharmaceutical Incorporated Company; and propyl chloride, Xi'an Libang Pharmacertical Company) .The patients received an ultrasonic bronchoscopy (the Olympus 290 electronic bronchoscopy system of Japanese Olympus Company) from the mouth, the glottis, through the trachea. The locations of the lymph nodes were initially determined according to preoperative imaging examination. The B-mode ultrasound was started and the image focus and depth of observation was adjusted after the ultrasonic water sac was filled, so that the whole target lymph nodes and the surrounding normal tissues were clearly displayed on the screen. the investigators observed multi sections, selected the largest layer of the target lymph node, and retained pictures.The ultrasound image characteristics were independently recorded by three skilled respiratory physicians. The results were discussed and judged until consensus was reached.

EBUS UE The B-mode was switched to the elastography mode. When the image was stable, it would be frozen and photographed. The observer judged the image type according to the color ratio of the image. Type 1: mainly non-blue (green and red); type 2: partly blue, partly non-blue (green and red); and type 3: mainly blue. Then, the strain rate ratios of normal tissue (green and red) and the hardest region (the deepest blue) in the target lymph node region were measured and recorded. In contrast to B-mode ultrasound lymph node images, the elastography images were taken out as region of interest (ROI) in Image J software. The ROI was converted into RGB encoding mode, and the blue part was extracted from the Metlab software by setting the difference between the B component and the R and G components. After that, the blue area to ROI area ratio was calculated. According to the blue area ratio, the following grading standard was used to evaluate each lymph node as follows. 1 point: over 80% of the section was non blue (green, yellow and red); 2 point: more than 50%, but less than 80% of the section was non-blue (green, yellow and red); 3 point: more than 50%, but less than 80% of the section was blue; and 4 point: over 80% of the section was blue.

EBUS-TBNA and Final Diagnosis After elastography, switch to the blood flow pattern, avoid the blood vessels, confirm the safe needle path to the target node and adjust the depth of the needle (Cook Ireland Limited Liability Company, Ireland). EBUS-TBNA was performed under the guidance of real-time ultrasound. Each target lymph node was punctured 3~4 times. All the histological and cytological specimens were analyzed by pathologists who were blinded to the elastography values. A positive diagnosis was confirmed by pathology and/or cytology, and all patients with negative results underwent thoracoscopic or open chest surgery and follow-up to confirm the benign and malignant lymph nodes.

Statistical Analysis All data statistics were analyzed by SPSS 22 (IBM, New York, USA) statistical software. The normal distribution data were described by mean and standard deviation, and the quantitative data were described by median (maximum and minimum), and the qualitative data were described by percentage. All the numerical variables were analyzed by one-way ANOVA, and the chi-square test was used for categorical variables. The difference was statistically significant when P<0.05. If the benign and malignant group values conformed to normal distribution and the variance was homogeneous, the independent sample t test was used, otherwise the nonparametric test (Mann-Whitney test) was utilized. ROC analysis was conducted to evaluate the diagnostic value of single characteristics and combined characteristics. The maximum Youden index was calculated to determine the optimal cut-off point of differential diagnosis of benign and malignant lymph nodes. The diagnostic accuracy, sensitivity, specificity, PPV and NPV of each meaningful characteristic and combined characteristics were calculated respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have enlarged intrathoracic lymph nodes(≥1cm) evaluated by chest enhanced CT and/or 18-FDG high uptake (SUV Max > 2.5) evaluated by 18-FDG PET-CT.
2. Patients who are willing to undergo electronic bronchoscopy and agreed to take TBNA and EBUS-TBNA for pathology.

Exclusion Criteria:

1. There is a contraindication of electronic bronchoscopy: activity of hemoptysis, hypertension and arrhythmia, recent myocardial infarction or unstable angina pectoris attacks, serious heart and lung dysfunction, bleeding tendency which cannot be corrected, serious obstruction of superior vena cava syndrome, suspected aortic aneurysm, multiple pulmonary bullous,the body condition is extremely exhaustion, the pregnant or lactation period women, the infected wound deferred, uncontrollable mental illness.
2. Patients who are not willing to accept electronic bronchoscopy.

Ages: 27 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The echo characteristic of the B-mode ultrasound of lymph nodes. | 10 minutes
  echo characteristic(hypoechoic or not hypoechoic, homogeneous or not)

SECONDARY OUTCOMES:
The shape of the B-mode ultrasound of lymph nodes. | 10 minutes
  shape (round or not)
The boundary of the B-mode ultrasound of lymph nodes. | 10 minutes
  boundary (clear or not）
The short diameter of the B-mode ultrasound of lymph nodes. | 10 minutes
  short diameter (millimeter，mm)
The image type of the elastography of lymph nodes. | 10 minutes
  image type ( Type 1: mainly non-blue (green and red);Type 2: partly blue, partly non-blue (green and red); Type 3: mainly blue )
The strain ratio of the elastography of lymph nodes. | 10 minutes
  strain ratio (ratio result)
The blue area ratio of the elastography of lymph nodes. | 15 minutes
  blue area ratio (The percentage of the number of blue pixels in the total number of pixels of the entire lymph node image,%)
The grading score of the elastography of lymph nodes. | 15 minutes
  grading score (The percentage of the number of specific color pixels in the total number of pixels of the entire lymph node image：1 point: over 80% of the section was non blue (green, yellow and red); 2 point: more than 50%, but less than 80% of the section was non-blue (green, yellow and red);3 point: more than 50%, but less than 80% of the section was blue; and 4 point: over 80% of the section was blue)

OTHER OUTCOMES:
The short diameter of the enhanced chest computed tomography of lymph nodes. | 30 minutes
  short diameter (millimeter，mm)
The texture of the enhanced chest computed tomography of lymph nodes. | 6 minutes
  texture (homogeneous or not)
The shape of the enhanced chest computed tomography of lymph nodes. | 6 minutes
  shape (round or not)
The boundary of the enhanced chest computed tomography of lymph nodes. | 6 minutes
  boundary (clear or not)
The mean CT value of the enhanced chest computed tomography of lymph nodes. | 6 minutes
  mean CT value（hounsfield unit，HU）

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gu, master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: Yes
We are willing to share data related to lymph nodes in patients who were involved in the study. Researchers can contact us via mail to get data information for further research if they would.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data is available now and in 3 years.
Access Criteria: Researchers who are involved in the study of ultrasound elastography with lymph nodes and contact contact us via mail until our agreement.

REFERENCES:
- [Background] Ophir J, Cespedes I, Ponnekanti H, Yazdi Y, Li X. Elastography: a quantitative method for imaging the elasticity of biological tissues. Ultrason Imaging. 1991 Apr;13(2):111-34. doi: 10.1177/016173469101300201. PMID 1858217
- [Background] Saftoiu A, Vilman P. Endoscopic ultrasound elastography-- a new imaging technique for the visualization of tissue elasticity distribution. J Gastrointestin Liver Dis. 2006 Jun;15(2):161-5. PMID 16802011
- [Background] Dietrich CF, Jenssen C, Herth FJ. Endobronchial ultrasound elastography. Endosc Ultrasound. 2016 Jul-Aug;5(4):233-8. doi: 10.4103/2303-9027.187866. PMID 27503154
- [Background] Dietrich CF, Saftoiu A, Jenssen C. Real time elastography endoscopic ultrasound (RTE-EUS), a comprehensive review. Eur J Radiol. 2014 Mar;83(3):405-14. doi: 10.1016/j.ejrad.2013.03.023. Epub 2013 May 1. PMID 23643030
- [Background] Zhou BG, Wang D, Ren WW, Li XL, He YP, Liu BJ, Wang Q, Chen SG, Alizad A, Xu HX. Value of shear wave arrival time contour display in shear wave elastography for breast masses diagnosis. Sci Rep. 2017 Aug 1;7(1):7036. doi: 10.1038/s41598-017-07389-0. PMID 28765627
- [Background] Zhang F, Zhao X, Han R, Du M, Li P, Ji X. Comparison of Acoustic Radiation Force Impulse Imaging and Strain Elastography in Differentiating Malignant From Benign Thyroid Nodules. J Ultrasound Med. 2017 Dec;36(12):2533-2543. doi: 10.1002/jum.14302. Epub 2017 Jun 24. PMID 28646602
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH. Shear-Wave Elastography for Detection of Prostate Cancer: A Systematic Review and Diagnostic Meta-Analysis. AJR Am J Roentgenol. 2017 Oct;209(4):806-814. doi: 10.2214/AJR.17.18056. Epub 2017 Aug 10. PMID 28796546
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Lim CK, Chung CL, Lin YT, Chang CH, Lai YC, Wang HC, Yu CJ. Transthoracic Ultrasound Elastography in Pulmonary Lesions and Diseases. Ultrasound Med Biol. 2017 Jan;43(1):145-152. doi: 10.1016/j.ultrasmedbio.2016.08.028. Epub 2016 Oct 12. PMID 27743728
- [Background] Izumo T, Sasada S, Chavez C, Matsumoto Y, Tsuchida T. Endobronchial ultrasound elastography in the diagnosis of mediastinal and hilar lymph nodes. Jpn J Clin Oncol. 2014 Oct;44(10):956-62. doi: 10.1093/jjco/hyu105. Epub 2014 Aug 13. PMID 25121724
- [Background] Furukawa MK, Kubota A, Hanamura H, Furukawa M. [Clinical application of real-time tissue elastography to head and neck cancer--evaluation of cervical lymph node metastasis with real-time tissue elastography]. Nihon Jibiinkoka Gakkai Kaiho. 2007 Jul;110(7):503-5. doi: 10.3950/jibiinkoka.110.503. Japanese. PMID 17695297
- [Background] Rusch VW, Asamura H, Watanabe H, Giroux DJ, Rami-Porta R, Goldstraw P; Members of IASLC Staging Committee. The IASLC lung cancer staging project: a proposal for a new international lymph node map in the forthcoming seventh edition of the TNM classification for lung cancer. J Thorac Oncol. 2009 May;4(5):568-77. doi: 10.1097/JTO.0b013e3181a0d82e. PMID 19357537